CLINICAL TRIAL: NCT02825732
Title: MEMORA-Caregiver : Risk Factors of Caregiver Burden Among Patients With Neurocognitive Disorders or Subjective Cognitive Complaint
Acronym: MEMORA
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL16_0437
Record Dates: First submitted 2016-07-04; First posted 2016-07-07 (Estimated); Last update posted 2016-07-11 (Estimated); Status verified 2016-07

CONDITIONS: Neurocognitive Disorders
Keywords: Alzheimer's disease or related disorder; Comorbidity; Charlson comorbidity index; Caregiver burden; Cohort; Dementia; Behavioral disorders; Functional dependency
MeSH Terms: conditions — Neurocognitive Disorders; Alzheimer Disease; Caregiver Burden; Dementia; Mental Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The investigators will investigate which patients' characteristics are associated with caregivers burden and its evolution for outpatients visiting a memory clinic, in particular how functional autonomy, behavioral and psychological symptoms as well as patients comorbidities can influence caregiver burden.

The study will be conducted among outpatients with progressive cognitive complaint followed in a Memory Clinic and their primary caregiver. The investigators hypothesis that caregivers experience a higher burden due to disease symptoms such as impairment of functional autonomy, behavioral and cognitive impairment, whatever the aetiology of the cognitive decline.

ELIGIBILITY:
Inclusion Criteria:

* patients with a cognitive complaint, either expressed by the patient or one of their relatives,
* patients at any stage of disease (cognitive complaint, mild cognitive impairment (MCI) or dementia),
* patients living in the community,
* patients having an informal caregiver who will complete the questionnaire to assess the caregiver burden.

Exclusion Criteria:

-

Ages: 50 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population includes a sample of consecutive dyads of patient-caregiver consulting a neurologist or a geriatrician for a cognitive complaint between November 2011 and December 2014 at the Memory Clinic of the Hospital Charpennes, Villeurbanne, France.
Sampling Method: Non-Probability Sample
Enrollment: 1300 (Actual)
Dates: Start 2011-11; Primary Completion 2014-12 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Evolution of caregiver burden | Two measured of the caregiver burden at baseline and at follow-up during current care, at 6 months to 12 months of follow-up.
  The caregiver burden change will be assessed using two repeated measures of the validated short version of the ZBI.

SECONDARY OUTCOMES:
Caregiver burden | The caregiver burden will be measured at baseline (Day 0)
  The caregivers burden will be assessed using the validated short version of the Zarit Burden Inventory (ZBI), which was previously developed for routine medical care. The score is noted as a continuous variable ranging from 0 (no burden) to 7 (higher burden). The questionnaire includes 7 questions for which the caregivers could answer "never", "sometimes" or "nearly always": Does the fact of caring for your relative lead to 1. Difficulties in your family life, 2. Difficulties in your relationship with friends, hobbies, or in your work, 3. An impact on your health, 4. Do you have the feeling of no longer recognizing your relative? 5. Are you concerned for the future of your relative? 6. Do you feel you need more help to take care of your relative? 7. Do you feel a burden in taking care of your relative? The questionnaire of ZBI will be sent at home and completed by the caregiver before the patient's consultation at the memory centre.

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Krolak-Salmon, Pr, Principal Investigator — Clinical and Research Memory Centre of Lyon (CMRR); Geriatrics Unit, Charpennes Hospital, University Hospital of Lyon, Villeurbanne, France - Clinical Research Centre (CRC) - VCF (Aging - Brain - Frailty), Charpennes Hospital, University Hospital of Lyon
Locations (1):
- Clinical and Research Memory Centre of Lyon (CMRR); Geriatrics Unit, Charpennes Hospital, University Hospital of Lyon, Villeurbanne, France - Clinical Research Centre (CRC) - VCF (Aging - Brain - Frailty), Charpennes Hospital, University Hospital of Lyon, Villeurbanne, France

REFERENCES:
- [Derived] Dauphinot V, Ravier A, Novais T, Delphin-Combe F, Mouchoux C, Krolak-Salmon P. Risk Factors of Caregiver Burden Evolution, for Patients With Subjective Cognitive Decline or Neurocognitive Disorders: A Longitudinal Analysis. J Am Med Dir Assoc. 2016 Nov 1;17(11):1037-1043. doi: 10.1016/j.jamda.2016.07.003. Epub 2016 Aug 26. PMID 27575984